CLINICAL TRIAL: NCT01875900
Title: Instructor-led Simulation Training Versus Self-directed Simulator Training During Simulated Neonatal Resuscitation - A Randomized Controlled Trial
Brief Title: Instructor-led Simulation Training Versus Self-directed Simulator Training During Simulated Neonatal Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Lukas P Mileder, MD, cand.med., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 25-399 ex 12/13
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Resuscitation; Neonatology
Keywords: neonatal resuscitation; video-assisted learning; self-directed training; simulation; simulation-based training; simulation-based medical education; objective structured clinical examination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video-assisted learning and self-directed training (Active Comparator): The Neonatal Resuscitation Program (NRP) digital video disc (DVD) will be provided for video study and a low-fidelity newborn manikin for self-directed resuscitation training (90 minutes training time, six students per group).
  Interventions: Other: Video-assisted learning and self-directed training
- Simulation-based neonatal resuscitation training (Experimental): Students will learn initial assessment of newborns and basic resuscitation skills and actively apply these skills during simulated clinical scenarios both with a low- and high-fidelity manikin (90 minutes training time, six students per group).
  Interventions: Other: Simulation-based neonatal resuscitation training

INTERVENTIONS:
Other: Video-assisted learning and self-directed training — The Neonatal Resuscitation Program (NRP) DVD will be provided for video study and a low-fidelity newborn manikin for self-directed resuscitation training (90 minutes training time, six students per group).
  Other Names: Visual learning and independent neonatal resuscitation training
  Arms: Video-assisted learning and self-directed training
Other: Simulation-based neonatal resuscitation training — Students will learn initial assessment of newborns and basic resuscitation skills and actively apply these skills during simulated clinical scenarios both with a low- and high-fidelity manikin (90 minutes training time, six students per group).
  Other Names: Instructor-led neonatal resuscitation training
  Arms: Simulation-based neonatal resuscitation training

SUMMARY:
Simulation-based training has been widely implemented in medical education. According to educational theories, simulation-based medical education (SBME) is associated with significant advantages, which has been investigated and proved by many studies. However, the value of SBME in comparison to other instructional methodologies remains largely unknown. Therefore, the aim of this study is to directly compare two instructional methods for neonatal resuscitation training.

ELIGIBILITY:
Inclusion Criteria:

* Fifth-year medical students prior to their mandatory OSCE
* Signing of informed consent

Exclusion Criteria:

* Refusal to participate in the study

The first two OSCEs in July and August will be part of a pilot study. The combined results of both examinations will be used for a sample size calculation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Neonatal resuscitation performance | Students will take part in an Objective Structured Clinical Examination (OSCE) within two weeks after having participated in the course.
  Students will perform neonatal resuscitation as part of an OSCE.

SECONDARY OUTCOMES:
Effectiveness of instructional methodology, success of OSCE preparation, transferability of skills into patient care | within two weeks
  Students will be asked to rate the subjective effectiveness of the respective instructional methodology, success of OSCE preparation, and transferability of skills into patient care using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmölzer, M.D., Ph.D., Study Chair — Division of Neonatology, Department of Pediatrics, Medical University of Graz, Austria; Department of Pediatrics, University of Alberta, Edmonton, Canada; Berndt Urlesberger, M.D., Study Chair — Division of Neonatology, Department of Pediatrics, Medical University of Graz, Austria; Ernst Eber, M.D., Study Chair — Respiratory and Allergic Disease Division , Department of Pediatrics, Medical University of Graz, Austria; Albrecht Schmidt, M.D., Study Chair — Division of Cardiology, Department of Internal Medicine, Medical University of Graz, Austria; Clinical Skills Center, Medical University of Graz, Austria
Locations (1):
- Clinical Skills Center, Medical University of Graz, Graz, Styria, Austria